CLINICAL TRIAL: NCT02116621
Title: N-of-1 Trials Using mHealth in Chronic Pain Aka PREEMPT (Personalized Research for Monitoring Pain Treatment)
Brief Title: N-of-1 Trials Using mHealth in Chronic Pain
Acronym: PREEMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 496804; R01NR001938 (NIH)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-03

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: Musculoskeletal pain; Chronic pain; Patient centered outcomes research; Physician patient relationship; Mobile applications
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trialist Intervention (Experimental): Clinician and patient set up N-of-1 trial 4-12 weeks in length to compare two treatments for chronic pain. Patient uses Trialist smartphone app to monitor pain and associated side effects daily throughout length of N-of-1 trial. After trial ends, the patient reviews graphical displays of N-of-1 trial results with clinician.
  Interventions: Behavioral: Trialist Intervention; Device: smartphone
- Control-Usual Care (No Intervention): Receive usual care from clinician for chronic pain, do not use Trialist smartphone app

INTERVENTIONS:
Behavioral: Trialist Intervention — Clinician and patient set up N-of-1 trial and patient uses Trialist smartphone app to answer daily questions about pain and associated side effects.
  Other Names: Trialist smartphone app; mobile health
  Arms: Trialist Intervention
Device: smartphone
  Arms: Trialist Intervention

SUMMARY:
Chronic musculoskeletal pain is an important problem, and treatments are often prescribed in a "trial and error" fashion. Clinicians prescribe a treatment to a patient and then wait and see if the treatment is successful. If the treatment is unsuccessful, they will try a different treatment. The disadvantage to this method is that it may take a long time to find a successful treatment.

The purpose of the PREEMPT Study is to test whether using a mobile phone application ("Trialist app") that allows patients and their health care providers to run personalized experiments comparing two pain treatments is more effective than usual care. Patients download the app, and working with their clinicians, set up a personalized trial that makes sense for them. Every day they answer questions to track levels of pain and side effects of treatment, such as fatigue and constipation. Once the personalized trial has ended, the responses to these daily questions on each treatment will be compared. During a regular clinic visit, the patient and the clinician will review visual displays of the results to facilitate treatment decision-making. Approximately 250 patients will be enrolled in the study. Half the patients will use the app and review results with the clinician, and half the patients will continue with their regular care (i.e., will not use the app). The two groups will be compared to see if using the app is successful in improving long term pain outcomes. The goal of the intervention using the Trialist app is to help patients engage actively and collaboratively with their clinicians and identify effective treatments more quickly.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (e.g., neck, back, extremities) operationalized as pain present for 6 weeks or more and a pain score of 4 or higher (on a 0-to-10 scale) on at least one of three items from the PEG pain scale
* Age 18-75 years
* Own web-enabled Android or iOS phone with data plan
* In judgment of treating clinician, pain potentially amenable to treatment with acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), low-dose opioids, a complementary/alternative treatment such as massage or meditation, or a simple combination of these treatments
* Ability to speak and read English

Exclusion Criteria:

* Treated with surgery, radiation or chemotherapy for cancer in past 5 years
* Other medical conditions that in clinician's judgment would limit life expectancy to less than 2 years or imperil patient safety
* Pregnant or breastfeeding
* Dementia, bipolar disorder, schizophrenia, active suicidality
* Current alcohol or prescription drug abuse; history of disruptive behavior
* Failed 5 or more analgesic medications because of lack of effectiveness or poor tolerability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Kravitz, MD, MSPH, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - Veteran's Administration-Northern California Health Care System, Mather, California
  - University of California, Davis Medical Center, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr C, Marois M, Sim I, Schmid CH, Wilsey B, Ward D, Duan N, Hays RD, Selsky J, Servadio J, Schwartz M, Dsouza C, Dhammi N, Holt Z, Baquero V, MacDonald S, Jerant A, Sprinkle R, Kravitz RL. The PREEMPT study - evaluating smartphone-assisted n-of-1 trials in patients with chronic pain: study protocol for a randomized controlled trial. Trials. 2015 Feb 27;16:67. doi: 10.1186/s13063-015-0590-8. PMID 25881274
- [Derived] Kravitz RL, Marois M, Sim I, Ward D, Kanekar SS, Yu A, Dounias P, Yang J, Wang Y, Schmid CH. Chronic pain treatment preferences change following participation in N-of-1 trials, but not always in the expected direction. J Clin Epidemiol. 2021 Nov;139:167-176. doi: 10.1016/j.jclinepi.2021.08.007. Epub 2021 Aug 14. PMID 34400254
- [Derived] Odineal DD, Marois MT, Ward D, Schmid CH, Cabrera R, Sim I, Wang Y, Wilsey B, Duan N, Henry SG, Kravitz RL. Effect of Mobile Device-Assisted N-of-1 Trial Participation on Analgesic Prescribing for Chronic Pain: Randomized Controlled Trial. J Gen Intern Med. 2020 Jan;35(1):102-111. doi: 10.1007/s11606-019-05303-0. Epub 2019 Aug 28. PMID 31463686
- [Derived] Kravitz RL, Schmid CH, Marois M, Wilsey B, Ward D, Hays RD, Duan N, Wang Y, MacDonald S, Jerant A, Servadio JL, Haddad D, Sim I. Effect of Mobile Device-Supported Single-Patient Multi-crossover Trials on Treatment of Chronic Musculoskeletal Pain: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1368-1377. doi: 10.1001/jamainternmed.2018.3981. PMID 30193253

RESULTS

PARTICIPANT FLOW:
Groups:
- Trialist Intervention: Clinician and patient set up N-of-1 trial 4-12 weeks in length to compare two treatments for chronic pain. Patient uses Trialist smartphone app to monitor pain and associated side effects daily throughout length of N-of-1 trial. After trial ends, the patient reviews graphical displays of N-of-1 trial results with clinician.
  Trialist Intervention: Clinician and patient set up N-of-1 trial and patient uses Trialist smartphone app to answer daily questions about pain and associated side effects.
  smartphone
Period: Baseline
Arm/Group | Trialist Intervention | Control-Usual Care
Started | 108 | 107
Completed Baseline Visit | 108 | 103
Completed Intervention Period | 95 | 103
Completed | 108 | 103
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4
Period: Three Month Follow-up
Arm/Group | Trialist Intervention | Control-Usual Care
Started | 108 | 103
Completed | 89 | 96
Not Completed | 19 | 7
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not complete follow-up survey | 14 | 4
Period: Six Month Follow-up
Arm/Group | Trialist Intervention | Control-Usual Care
Started | 103 (Patients who didn't complete 3mo survey but didn't drop from study were contacted for 6mo follow-up.) | 100 (Patients who didn't complete 3mo survey but didn't drop from study were contacted for 6mo follow-up)
Completed | 99 | 97
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Did not complete follow-up survey | 1 | 1
Period: Twelve Month Follow-up
Arm/Group | Trialist Intervention | Control-Usual Care
Started | 100 (Patients who didn't complete 6mo survey but didn't drop from study were contacted for 12mo follow-up) | 98 (Patients who didn't complete 6mo survey but didn't drop from study were contacted for 12mo follow-up)
Completed | 84 | 86
Not Completed | 16 | 12
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not complete follow-up survey | 1 | 3
Not completed — Enrolled within 12 months of study end | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trialist Intervention | Control-Usual Care | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.8) | 55.6 (11.5) | 55.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 58 | 55 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 8 | 24
  Not Hispanic or Latino | 91 | 95 | 186
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 75 | 80 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 8 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 107 | 215
Pain interference [Mean (Standard Deviation); unit: units on a scale] — Pain interference measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item short form which measures self-reported consequences of pain on relevant aspects of one's life. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain interference scores range from 0 - 100. For pain interference, higher scores indicate greater pain interference.
  units on a scale | 64.0 (5.9) | 64.7 (5.8) | 64.3 (5.8)
Pain intensity [Mean (Standard Deviation); unit: units on a scale] — Pain intensity measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 3a short form which measures self-reported estimate of how much a person hurts. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain intensity scores range from 0 - 100. For pain intensity, higher scores indicate greater pain intensity.
  units on a scale | 53.5 (5.4) | 53.8 (5.1) | 53.7 (5.2)
Global physical health [Mean (Standard Deviation); unit: units on a scale] — Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale, representing physical and mental health components. Global physical health measures overall physical health, physical function, pain and fatigue. The final physical health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Physical global health scores range from 0 - 100, and higher scores indicate better physical health.
  units on a scale | 42.5 (6.8) | 40.6 (5.5) | 41.6 (6.2)
Global mental health [Mean (Standard Deviation); unit: units on a scale] — Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale, representing physical and mental health components. Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. The final mental health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Global mental health scores range from 0 - 100, and higher scores indicate better mental health.
  units on a scale | 44.9 (9.1) | 43.2 (7.9) | 44.1 (8.6)
Analgesic adherence (overuse) [Mean (Standard Deviation); unit: units on a scale] — Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications. Two questions comprised a subscale assessing overuse of medications. Overuse scores range from 0 - 100. Higher scores indicate greater adherence and less overuse of medications.
  units on a scale | 90.2 (12.4) | 89.4 (13.4) | 89.8 (12.9)
Analgesic adherence (underuse) [Mean (Standard Deviation); unit: units on a scale] — Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications. Two questions comprised a subscale assessing underuse of medications. Underuse scores range from 0-100. Higher scores indicate greater adherence and less underuse of medication.
  units on a scale | 75.2 (22.3) | 75.6 (24.6) | 75.4 (23.4)
Trust in clinician [Mean (Standard Deviation); unit: units on a scale] — Patient trust in physician measured with 11-item Trust in Physician Scale to assess the quality of the patient-clinician relationship. Trust in physician scores range from 0 - 100. Higher scores indicate greater patient trust in the clinician providing pain treatment.
  units on a scale | 76.8 (15.8) | 75.3 (17.1) | 76.1 (16.4)
Satisfaction with pain information [Mean (Standard Deviation); unit: units on a scale] — The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction, creating three subscales. Satisfaction with pain information is a subscale that includes 5 questions assessing information about pain and its treatment. Satisfaction with pain information range from 0-100. Higher scores indicate greater patient satisfaction with information received about pain and treatment for pain.
  units on a scale | 50.5 (38.8) | 50.7 (37.8) | 50.6 (38.2)
Satisfaction with medical care [Mean (Standard Deviation); unit: units on a scale] — The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction, creating three subscales. Satisfaction with medical care is a subscale that includes 5 questions assessing medical care for pain. Satisfaction with medical care scores range from 0 - 100. Higher scores indicate greater patient satisfaction with medical care.
  units on a scale | 84.7 (15.7) | 79.5 (19.2) | 82.2 (17.7)
Satisfaction with pain medication [Mean (Standard Deviation); unit: units on a scale] — The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction, creating three subscales. Satisfaction with current pain medication is a subscale that includes 8 questions assessing current pain medications. Satisfaction with pain medication scores range from 0-100. Higher scores indicate greater patient satisfaction with current pain medications.
  units on a scale | 65.2 (22.1) | 63.4 (23.6) | 64.4 (22.8)
Medication related shared decision making [Mean (Standard Deviation); unit: units on a scale] — Four questions from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) survey assessed patient-provider discussions on starting/stopping medications and comprise medication related shared decision making. Scores were computed only for patients who reported discussing medications with their clinician in the past 12 months. Medication related shared decision making scores range from 0-100. Higher scores indicate more shared decision making.
  units on a scale | 74.3 (23.8) | 75.0 (24.3) | 74.6 (23.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain-related Interference on the Patient Reported Outcomes Measurement Information System (PROMIS) Scale at 26 Weeks
Description: Pain interference measured with Patient Reported Outcomes Measurement Information System (PROMIS) Scale 8-item short form at baseline and 26 weeks which measures self-reported consequences of pain on relevant aspects of one's life. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain interference scores range from 0 - 100. For pain interference, higher scores indicate greater pain interference. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain interference.
Time Frame: baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -3.22 [-4.31 to -2.13] | -1.85 [-2.96 to -0.75]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -1.36, 95% CI 2-sided [-2.91 to 0.19] — Adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control) from baseline to 26 weeks

2. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up in Pain-related Interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale
Description: Pain-related Interference measured with Patient-Reported Outcomes Measurement Information System (PROMIS) scale 8-item short form at baseline, 13 weeks, 26 weeks, and 52 weeks which measures self-reported consequences of pain on relevant aspects of one's life. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain interference scores range from 0 - 100. For pain interference, higher scores indicate greater pain interference. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain interference.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: Longitudinal analysis at baseline, 13, 26 and 52 weeks; numbers reported are adjusted means from a mixed effect Gaussian model using time, treatment and time*treatment interaction as fixed effects and clinician and patient as random effects.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | -2.70 [-3.83 to -1.57] | -1.91 [-3.02 to -0.81]
  Change from baseline to 26 weeks | -3.22 [-4.31 to -2.13] | -1.85 [-2.96 to -0.75]
  Change from baseline to 52 weeks | -2.67 [-3.82 to -1.52] | -2.83 [-3.98 to -1.68]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.21, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: -0.79 (-2.37 to 0.80); baseline to 26 weeks: -1.36 (-2.91 to 0.19); baseline to 52 weeks: 0.16 (-1.47 to 1.79)

3. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up in Pain Intensity on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale
Description: Pain intensity measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 3a short form at baseline, 13 weeks, 26 weeks, and 52 weeks which measures self-reported estimate of how much a person hurts. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain intensity scores range from 0 - 100. For pain intensity, higher scores indicate greater pain intensity. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain intensity.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | -1.60 [-2.67 to -0.54] | -1.92 [-2.96 to -0.87]
  Change from baseline to 26 weeks | -2.86 [-3.89 to -1.83] | -1.46 [-2.50 to -0.41]
  Change from baseline to 52 weeks | -3.00 [-4.08 to -1.91] | -1.76 [-2.85 to -0.67]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.06, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 0.31 (-1.18 to 1.81); baseline to 26 weeks: -1.41 (-2.87 to 0.06); baseline to 52 weeks: -1.24 (-2.77 to 0.30)

4. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up on the Patient-Reported Outcomes Measurement Information System (PROMIS) MENTAL Global Health Scale
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline, 13 weeks, 26 weeks, and 52 weeks, representing physical and mental health components. Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. The final mental health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Global mental health scores range from 0 - 100, and higher scores indicate better mental health. Data table measures show change over time with positive numbers indicating improvement in global mental health and negative numbers indicating declines in global mental health.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | -0.35 [-1.71 to 1.00] | 0.30 [-1.02 to 1.63]
  Change from baseline to 26 weeks | 0.21 [-1.09 to 1.52] | -0.72 [-2.04 to 0.60]
  Change from baseline to 52 weeks | 0.36 [-1.01 to 1.74] | -0.39 [-1.76 to 0.98]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.35, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks:-0.66 (-2.55 to 1.24); baseline to 26 weeks: 0.93 (-0.92 to 2.79); baseline to 52 weeks: 0.76 (-1.19 to 2.70)

5. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up on the Patient-Reported Outcomes Measurement Information System (PROMIS) PHYSICAL Global Health Scale
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline, 13 weeks, 26 weeks, 52 weeks, representing physical and mental health components. Global physical health measures overall physical health, physical function, pain and fatigue. The final physical health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Physical global health scores range from 0 - 100, and higher scores indicate better physical health. Data table measures show change over time with positive numbers indicating improvement in global physical health and negative numbers indicating declines in global physical health.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | 0.73 [-0.21 to 1.67] | 0.44 [-0.48 to 1.35]
  Change from baseline to 26 weeks | 0.13 [-0.77 to 1.03] | 0.30 [-0.61 to 1.21]
  Change from baseline to 52 weeks | 0.16 [-0.79 to 1.12] | 0.42 [-0.53 to 1.37]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.86, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 0.30 (-1.01 to 1.61); baseline to 26 weeks: -0.17 (-1.45 to 1.12); baseline to 52 weeks: -0.26 (-1.61 to 1.09)

6. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up in Analgesic Adherence (Overuse) on the Pain Medication in Primary Care Patient Questionnaire
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline, 13 weeks, 26 weeks, 52 weeks. Two questions comprised a subscale assessing overuse of medications. Overuse scores range from 0 - 100. Higher scores indicate greater adherence and less overuse of medications. Data table measures show change over time with positive numbers indicating greater adherence (less overuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | 1.40 [-1.18 to 3.98] | 0.35 [-2.15 to 2.85]
  Change from baseline to 26 weeks | 1.77 [-0.75 to 4.30] | -0.13 [-2.64 to 2.39]
  Change from baseline to 52 weeks | 1.61 [-1.02 to 4.24] | 1.53 [-1.06 to 4.12]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.70, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 1.05 (-2.54 to 4.64); baseline to 26 weeks: 1.90 (-1.66 to 5.47); baseline to 52 weeks: 0.08 (-3.61 to 3.77)

7. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up in Analgesic Adherence (Underuse) on the Pain Medication in Primary Care Patient Questionnaire
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline, 13 weeks, 26 weeks, 52 weeks. Two questions comprised a subscale assessing underuse of medications. Underuse scores range from 0-100. Higher scores indicate greater adherence and less underuse of medication. Data table measures show change over time with positive numbers indicating greater adherence (less underuse of medications) and negative numbers indicating less adherence.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | 2.53 [-2.46 to 7.52] | -1.71 [-6.56 to 3.15]
  Change from baseline to 26 weeks | 1.88 [-3.00 to 6.76] | -2.76 [-7.63 to 2.11]
  Change from baseline to 52 weeks | -3.53 [-8.62 to 1.56] | -1.62 [-6.66 to 3.42]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.20, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 4.24 (-2.73 to 11.20); baseline to 26 weeks: 4.64 (-2.25 to 11.54); baseline to 52 weeks: -1.91 (-9.07 to 5.26)

8. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up in Patient-provider Relationship on the Trust in Physician Scale
Description: Patient trust in physician measured with 11-item Trust in Physician Scale at baseline, 13 weeks, 26 weeks, and 52 weeks to assess the quality of the patient-clinician relationship. Trust in physician scores range from 0 - 100. Higher scores indicate greater patient trust in the clinician providing pain treatment. Data table measures show change over time with positive numbers indicating increases in trust and negative numbers indicating declines in trust.
Time Frame: baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | -2.49 [-5.44 to 0.46] | -4.25 [-7.13 to -1.36]
  Change from baseline to 26 weeks | -2.30 [-5.14 to 0.54] | -4.84 [-7.73 to -1.96]
  Change from baseline to 52 weeks | -4.00 [-7.00 to -0.99] | -5.53 [-8.52 to -2.54]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.66, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 1.76 (-2.37 to 5.89); baseline to 26 weeks: 2.55 (-1.50 to 6.60); baseline to 52 weeks: 1.53 (-2.70 to 5.77)

9. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up on the Pain Treatment Satisfaction Scale (PTSS) -Satisfaction With Pain Information
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline, 13 weeks, 26 weeks, and 52 weeks, creating three subscales. Satisfaction with pain information is a subscale that includes 5 questions assessing information about pain and its treatment. Satisfaction with pain information range from 0-100. Higher scores indicate greater patient satisfaction with information received about pain and treatment for pain. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain information and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | 4.41 [-3.18 to 12.00] | -3.36 [-10.84 to 4.11]
  Change from baseline to 26 weeks | 11.28 [3.95 to 18.61] | 3.99 [-3.47 to 11.45]
  Change from baseline to 52 weeks | 9.02 [1.28 to 16.76] | 4.89 [-2.84 to 12.63]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.44, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 7.77 (-2.87 to 18.42); baseline to 26 weeks: 7.29 (-3.16 to 17.75); baseline to 52 weeks: 4.13 (-6.81 to 15.07)

10. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up on the Pain Treatment Satisfaction Scale (PTSS) -Satisfaction With Medical Care
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline, 13 weeks, 26 weeks, 52 weeks, creating three subscales. Satisfaction with medical care is a subscale that includes 5 questions assessing medical care for pain. Satisfaction with medical care scores range from 0 - 100. Higher scores indicate greater patient satisfaction with medical care. Data table measures show change over time with positive numbers indicating increases in satisfaction with medical care and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | -4.00 [-7.56 to -0.44] | -6.15 [-9.64 to -2.66]
  Change from baseline to 26 weeks | -2.26 [-5.68 to 1.17] | -5.57 [-9.04 to -2.09]
  Change from baseline to 52 weeks | -4.52 [-8.13 to -0.90] | -5.51 [-9.12 to -1.91]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.58, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 2.15 (-2.84 to 7.13); baseline to 26 weeks: 3.31 (-1.57 to 8.19); baseline to 52 weeks: 1.00 (-4.11 to 6.11)

11. Secondary Outcome: Longitudinal Change From Baseline up to 52 Weeks Follow-up on the Pain Treatment Satisfaction Scale (PTSS) -Satisfaction With Pain Medication
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline, 13 weeks, 26 weeks, 52 weeks, creating three subscales. Satisfaction with current pain medication is a subscale that includes 8 questions assessing current pain medications. Satisfaction with pain medication scores range from 0-100. Higher scores indicate greater patient satisfaction with current pain medications. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain medications and negative numbers indicating declines in satisfaction with pain medications.
Time Frame: Baseline, 13 weeks, 26 weeks, 52 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale
  Change from baseline to 13 weeks | 1.46 [-2.93 to 5.86] | -0.34 [-4.73 to 4.05]
  Change from baseline to 26 weeks | -0.18 [-4.44 to 4.08] | 1.39 [-2.99 to 5.77]
  Change from baseline to 52 weeks | 0.77 [-3.72 to 5.25] | -0.34 [-4.87 to 4.19]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.73, Mixed Models Analysis; Longitudinal analysis adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control). Baseline to 13 weeks: 1.81 (-4.41 to 8.02); baseline to 26 weeks: -1.57 (-7.68 to 4.54); baseline to 52 weeks: 1.11 (-5.27 to 7.48)

12. Other Pre Specified Outcome: Change From Baseline in Pain Intensity on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale at 26 Weeks
Description: Pain intensity measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 3a short form at baseline and 26 weeks, which measures self-reported estimate of how much a person hurts. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain intensity scores range from 0 - 100. For pain intensity, higher scores indicate greater pain intensity. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain intensity.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.86 [-3.89 to -1.83] | -1.46 [-2.50 to -0.41]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -1.41, 95% CI 2-sided [-2.87 to 0.06] — [estimate comment as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) MENTAL Global Health Scale at 26 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 26 weeks, representing physical and mental health components. Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. The final mental health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Global mental health scores range from 0 - 100, and higher scores indicate better mental health. Data table measures show change over time with positive numbers indicating improvement in global mental health and negative numbers indicating declines in global mental health.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.21 [-1.09 to 1.52] | -0.72 [-2.04 to 0.60]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.93, 95% CI 2-sided [-0.92 to 2.79]; Adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control) from baseline to 26 weeks

14. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) PHYSICAL Global Health Scale at 26 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 26 weeks, representing physical and mental health components. Global physical health measures overall physical health, physical function, pain and fatigue. The final physical health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Physical global health scores range from 0 - 100, and higher scores indicate better physical health. Data table measures show change over time with positive numbers indicating improvement in global physical health and negative numbers indicating declines in global physical health.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.13 [-0.77 to 1.03] | 0.30 [-0.61 to 1.21]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -0.17, 95% CI 2-sided [-1.45 to 1.12]; [other analysis details as in outcome 13, analysis 1]

15. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Overuse) on the Pain Medication in Primary Care Patient Questionnaire at 26 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 26 weeks. Two questions comprised a subscale assessing overuse of medications. Overuse scores range from 0 - 100. Higher scores indicate greater adherence and less overuse of medications. Data table measures show change over time with positive numbers indicating greater adherence (less overuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 1.77 [-0.75 to 4.30] | -0.13 [-2.64 to 2.39]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.90, 95% CI 2-sided [-1.66 to 5.47]; [other analysis details as in outcome 13, analysis 1]

16. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Underuse) on the Pain Medication in Primary Care Patient Questionnaire at 26 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 26 weeks. Two questions comprised a subscale assessing underuse of medications. Underuse scores range from 0-100. Higher scores indicate greater adherence and less underuse of medication. Data table measures show change over time with positive numbers indicating greater adherence (less underuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 1.88 [-3.00 to 6.76] | -2.76 [-7.63 to 2.11]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 4.64, 95% CI 2-sided [-2.25 to 11.54]; [other analysis details as in outcome 13, analysis 1]

17. Other Pre Specified Outcome: Change From Baseline in Patient-provider Relationship on the Trust in Physician Scale at 26 Weeks
Description: Patient trust in physician measured with 11-item Trust in Physician Scale at baseline and 26 weeks to assess the quality of the patient-clinician relationship. Trust in physician scores range from 0 - 100. Higher scores indicate greater patient trust in the clinician providing pain treatment. Data table measures show change over time with positive numbers indicating increases in trust and negative numbers indicating declines in trust.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.30 [-5.14 to 0.54] | -4.84 [-7.73 to -1.96]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 2.55, 95% CI 2-sided [-1.50 to 6.60]; [other analysis details as in outcome 13, analysis 1]

18. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Information at 26 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 26 weeks, creating three subscales. Satisfaction with pain information is a subscale that includes 5 questions assessing information about pain and its treatment. Satisfaction with pain information range from 0-100. Higher scores indicate greater patient satisfaction with information received about pain and treatment for pain. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain information and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 11.28 [3.95 to 18.61] | 3.99 [-3.47 to 11.45]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 7.29, 95% CI 2-sided [-3.16 to 17.75]; [other analysis details as in outcome 13, analysis 1]

19. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Medical Care at 26 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 26 weeks, creating three subscales. Satisfaction with medical care is a subscale that includes 5 questions assessing medical care for pain. Satisfaction with medical care scores range from 0 - 100. Higher scores indicate greater patient satisfaction with medical care. Data table measures show change over time with positive numbers indicating increases in satisfaction with medical care and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.26 [-5.68 to 1.17] | -5.57 [-9.04 to -2.09]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 3.31, 95% CI 2-sided [-1.57 to 8.19]; [other analysis details as in outcome 13, analysis 1]

20. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Medication at 26 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 26 weeks, creating three subscales. Satisfaction with current pain medication is a subscale that includes 8 questions assessing current pain medications. Satisfaction with pain medication scores range from 0-100. Higher scores indicate greater patient satisfaction with current pain medications. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain medications and negative numbers indicating declines in satisfaction with pain medications.
Time Frame: Baseline, 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -0.18 [-4.44 to 4.08] | 1.39 [-2.99 to 5.77]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -1.57, 95% CI 2-sided [-7.68 to 4.54]; [other analysis details as in outcome 13, analysis 1]

21. Other Pre Specified Outcome: Change From Baseline in Participatory Decision-making on the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surveys at 26 Weeks
Description: Four questions from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) survey assessed patient-provider discussions on starting/stopping medications and comprise medication related shared decision making. Scores were computed only for patients who reported discussing medications with their clinician in the past 12 months. Medication related shared decision making scores range from 0-100. Higher scores indicate more shared decision making.
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 62 | 45
units on a scale | 79.6 [74.9 to 84.3] | 67.7 [58.7 to 76.7]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.01, Regression, Linear; Mean Difference (Final Values) = 11.9, 95% CI 2-sided [2.59 to 21.24]

22. Other Pre Specified Outcome: Change From Baseline in Pain-related Interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale at 13 Weeks
Description: Pain-related interference measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item short form at baseline and 13 weeks which measures self-reported consequences of pain on relevant aspects of one's life. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain interference scores range from 0 - 100. For pain interference, higher scores indicate greater pain interference. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain interference.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.70 [-3.83 to -1.57] | -1.91 [-3.02 to -0.81]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -0.79, 95% CI 2-sided [-2.37 to 0.80] — Adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control) from baseline to 13 weeks

23. Other Pre Specified Outcome: Change From Baseline in Pain Intensity on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale at 13 Weeks
Description: Pain intensity measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 3a short form at baseline and 13 weeks, which measures self-reported estimate of how much a person hurts. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain intensity scores range from 0 - 100. For pain intensity, higher scores indicate greater pain intensity. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain intensity.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -1.60 [-2.67 to -0.54] | -1.92 [-2.96 to -0.87]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.31, 95% CI 2-sided [-1.18 to 1.81] — [estimate comment as in outcome 22, analysis 1]

24. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) PHYSICAL Global Health Scale at 13 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 13 weeks, representing physical and mental health components. Global physical health measures overall physical health, physical function, pain and fatigue. The final physical health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Physical global health scores range from 0 - 100, and higher scores indicate better physical health. Data table measures show change over time with positive numbers indicating improvement in global physical health and negative numbers indicating declines in global physical health.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.73 [-0.21 to 1.67] | 0.44 [-0.48 to 1.35]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.30, 95% CI 2-sided [-1.01 to 1.61] — [estimate comment as in outcome 22, analysis 1]

25. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) MENTAL Global Health Scale at 13 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 13 weeks, representing physical and mental health components. Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. The final mental health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Global mental health scores range from 0 - 100, and higher scores indicate better mental health. Data table measures show change over time with positive numbers indicating improvement in global mental health and negative numbers indicating declines in global mental health.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -0.35 [-1.71 to 1.00] | 0.30 [-1.02 to 1.63]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -0.66, 95% CI 2-sided [-2.55 to 1.24] — [estimate comment as in outcome 22, analysis 1]

26. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Overuse) on the Pain Medication in Primary Care Patient Questionnaire at 13 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 13 weeks. Two questions comprised a subscale assessing overuse of medications. Overuse scores range from 0 - 100. Higher scores indicate greater adherence and less overuse of medications. Data table measures show change over time with positive numbers indicating greater adherence (less overuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 1.40 [-1.18 to 3.98] | 0.35 [-2.15 to 2.85]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.05, 95% CI 2-sided [-2.54 to 4.64] — [estimate comment as in outcome 22, analysis 1]

27. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Underuse) on the Pain Medication in Primary Care Patient Questionnaire at 13 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 13 weeks. Two questions comprised a subscale assessing underuse of medications. Underuse scores range from 0-100. Higher scores indicate greater adherence and less underuse of medication. Data table measures show change over time with positive numbers indicating greater adherence (less underuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 2.53 [-2.46 to 7.52] | -1.71 [-6.56 to 3.15]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 4.24, 95% CI 2-sided [-2.73 to 11.20] — [estimate comment as in outcome 22, analysis 1]

28. Other Pre Specified Outcome: Change From Baseline in Patient-provider Relationship on the Trust in Physician Scale at 13 Weeks
Description: Patient trust in physician measured with 11-item Trust in Physician Scale at baseline and 13 weeks to assess the quality of the patient-clinician relationship. Trust in physician scores range from 0 - 100. Higher scores indicate greater patient trust in the clinician providing pain treatment. Data table measures show change over time with positive numbers indicating increases in trust and negative numbers indicating declines in trust.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.49 [-5.44 to 0.46] | -4.25 [-7.13 to -1.36]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.76, 95% CI 2-sided [-2.37 to 5.89] — [estimate comment as in outcome 22, analysis 1]

29. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Information at 13 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 13 weeks, creating three subscales. Satisfaction with pain information is a subscale that includes 5 questions assessing information about pain and its treatment. Satisfaction with pain information range from 0-100. Higher scores indicate greater patient satisfaction with information received about pain and treatment for pain. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain information and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 4.41 [-3.18 to 12.00] | -3.36 [-10.84 to 4.11]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 7.77, 95% CI 2-sided [-2.87 to 18.42] — [estimate comment as in outcome 22, analysis 1]

30. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Medical Care at 13 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 13 weeks, creating three subscales. Satisfaction with medical care is a subscale that includes 5 questions assessing medical care for pain. Satisfaction with medical care scores range from 0 - 100. Higher scores indicate greater patient satisfaction with medical care. Data table measures show change over time with positive numbers indicating increases in satisfaction with medical care and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -4.00 [-7.56 to -0.44] | -6.15 [-9.64 to -2.66]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 2.15, 95% CI 2-sided [-2.84 to 7.13] — [estimate comment as in outcome 22, analysis 1]

31. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Medication at 13 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 13 weeks, creating three subscales. Satisfaction with current pain medication is a subscale that includes 8 questions assessing current pain medications. Satisfaction with pain medication scores range from 0-100. Higher scores indicate greater patient satisfaction with current pain medications. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain medications and negative numbers indicating declines in satisfaction with pain medications.
Time Frame: Baseline, 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 1.46 [-2.93 to 5.86] | -0.34 [-4.73 to 4.05]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.81, 95% CI 2-sided [-4.41 to 8.02] — [estimate comment as in outcome 22, analysis 1]

32. Other Pre Specified Outcome: Change From Baseline in Pain-related Interference on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale at 52 Weeks
Description: Pain-related interference measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item short form at baseline and 52 weeks which measures self-reported consequences of pain on relevant aspects of one's life. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain interference scores range from 0 - 100. For pain interference, higher scores indicate greater pain interference. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain interference.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -2.67 [-3.82 to -1.52] | -2.83 [-3.98 to -1.68]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.16, 95% CI 2-sided [-1.47 to 1.79] — Adjusted difference in differences using mixed effects Gaussian model (Trialist intervention - control) from baseline to 52 weeks

33. Other Pre Specified Outcome: Change From Baseline in Pain Intensity on the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale at 52 Weeks
Description: Pain intensity measured with Patient-Reported Outcomes Measurement Information System (PROMIS) 3a short form at baseline and 52 weeks, which measures self-reported estimate of how much a person hurts. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Pain intensity scores range from 0 - 100. For pain intensity, higher scores indicate greater pain intensity. Data table measures show change over time with negative numbers indicating improvement (decreases) and positive numbers indicating increases in pain intensity.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -3.00 [-4.08 to -1.91] | -1.76 [-2.85 to -0.67]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -1.24, 95% CI 2-sided [-2.77 to 0.30] — [estimate comment as in outcome 32, analysis 1]

34. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) PHYSICAL Global Health Scale at 52 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 52 weeks, representing physical and mental health components. Global physical health measures overall physical health, physical function, pain and fatigue. The final physical health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Physical global health scores range from 0 - 100, and higher scores indicate better physical health. Data table measures show change over time with positive numbers indicating improvement in global physical health and negative numbers indicating declines in global physical health.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.16 [-0.79 to 1.12] | 0.42 [-0.53 to 1.37]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -0.26, 95% CI 2-sided [-1.61 to 1.09] — [estimate comment as in outcome 32, analysis 1]

35. Other Pre Specified Outcome: Change From Baseline on the Patient-Reported Outcomes Measurement Information System (PROMIS) MENTAL Global Health Scale at 52 Weeks
Description: Global health measured with 10 item Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health scale at baseline and 52 weeks, representing physical and mental health components. Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. The final mental health score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Global mental health scores range from 0 - 100, and higher scores indicate better mental health. Data table measures show change over time with positive numbers indicating improvement in global mental health and negative numbers indicating declines in global mental health.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.36 [-1.01 to 1.74] | -0.39 [-1.76 to 0.98]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.76, 95% CI 2-sided [-1.19 to 2.70] — [estimate comment as in outcome 32, analysis 1]

36. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Overuse) on the Pain Medication in Primary Care Patient Questionnaire at 52 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 52 weeks. Two questions comprised a subscale assessing overuse of medications. Overuse scores range from 0 - 100. Higher scores indicate greater adherence and less overuse of medications. Data table measures show change over time with positive numbers indicating greater adherence (less overuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 1.61 [-1.02 to 4.24] | 1.53 [-1.06 to 4.12]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 0.08, 95% CI 2-sided [-3.61 to 3.77] — [estimate comment as in outcome 32, analysis 1]

37. Other Pre Specified Outcome: Change From Baseline in Analgesic Adherence (Underuse) on the Pain Medication in Primary Care Patient Questionnaire at 52 Weeks
Description: Four questions from the Pain Medication in Primary Care Patient Questionnaire measured adherence to medications at baseline and 52 weeks. Two questions comprised a subscale assessing underuse of medications. Underuse scores range from 0-100. Higher scores indicate greater adherence and less underuse of medication. Data table measures show change over time with positive numbers indicating greater adherence (less underuse of medications) and negative numbers indicating less adherence.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -3.53 [-8.62 to 1.56] | -1.62 [-6.66 to 3.42]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = -1.91, 95% CI 2-sided [-9.07 to 5.26] — [estimate comment as in outcome 32, analysis 1]

38. Other Pre Specified Outcome: Change From Baseline in Patient-provider Relationship on the Trust in Physician Scale at 52 Weeks
Description: Patient trust in physician measured with 11-item Trust in Physician Scale at baseline and 52 weeks to assess the quality of the patient-clinician relationship. Trust in physician scores range from 0 - 100. Higher scores indicate greater patient trust in the clinician providing pain treatment. Data table measures show change over time with positive numbers indicating increases in trust and negative numbers indicating declines in trust.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -4.00 [-7.00 to -0.99] | -5.53 [-8.52 to -2.54]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.53, 95% CI 2-sided [-2.70 to 5.77] — [estimate comment as in outcome 32, analysis 1]

39. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Information at 52 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 52 weeks, creating three subscales. Satisfaction with pain information is a subscale that includes 5 questions assessing information about pain and its treatment. Satisfaction with pain information range from 0-100. Higher scores indicate greater patient satisfaction with information received about pain and treatment for pain. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain information and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 9.02 [1.28 to 16.76] | 4.89 [-2.84 to 12.63]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 4.13, 95% CI 2-sided [-6.81 to 15.07] — [estimate comment as in outcome 32, analysis 1]

40. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Medical Care at 52 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 52 weeks, creating three subscales. Satisfaction with medical care is a subscale that includes 5 questions assessing medical care for pain. Satisfaction with medical care scores range from 0 - 100. Higher scores indicate greater patient satisfaction with medical care. Data table measures show change over time with positive numbers indicating increases in satisfaction with medical care and negative numbers indicating declines in patient satisfaction.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | -4.52 [-8.13 to -0.90] | -5.51 [-9.12 to -1.91]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.00, 95% CI 2-sided [-4.11 to 6.11] — [estimate comment as in outcome 32, analysis 1]

41. Other Pre Specified Outcome: Change From Baseline on the Pain Treatment Satisfaction Scale (PTSS) - Satisfaction With Pain Medication at 52 Weeks
Description: The Pain Treatment Satisfaction Scale consists of 18 items assessing patient satisfaction at baseline and 52 weeks, creating three subscales. Satisfaction with current pain medication is a subscale that includes 8 questions assessing current pain medications. Satisfaction with pain medication scores range from 0-100. Higher scores indicate greater patient satisfaction with current pain medications. Data table measures show change over time with positive numbers indicating increases in satisfaction with pain medications and negative numbers indicating declines in satisfaction with pain medications.
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 108 | 103
units on a scale | 0.77 [-3.72 to 5.25] | -0.34 [-4.87 to 4.19]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; Adjusted difference in differences = 1.11, 95% CI 2-sided [-5.27 to 7.48] — [estimate comment as in outcome 32, analysis 1]

42. Other Pre Specified Outcome: Change From Baseline in Participatory Decision-making on the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surveys at 52 Weeks
Description: as for outcome 21
Time Frame: Baseline, 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trialist Intervention | Control-Usual Care
Number analyzed (Participants) | 48 | 51
units on a scale | 74.8 [69.0 to 80.6] | 65.4 [57.7 to 73.0]
Statistical Analysis 1: Comparison: Trialist Intervention vs Control-Usual Care; Test type: Superiority; p = 0.054, Regression, Linear; Mean Difference (Final Values) = 9.41, 95% CI 2-sided [-0.15 to 18.96]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Trialist Intervention | Control-Usual Care
All-Cause Mortality (participants affected / at risk) | 1/108 | 1/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107
Other Adverse Events (participants affected / at risk) | 0/108 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT02116621/Prot_SAP_000.pdf